CLINICAL TRIAL: NCT06268171
Title: Ultrasound Assessment of Rectus Femoris Cross-sectionnal Area Following Lung Transplantation
Acronym: EchoSS-TP
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_0214; 2023-A02390-45 (Other: ANSM)
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Lung Transplant; Physiotherapy; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 61 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: transplant patients with ultrasound measurement of the cross-sectional area of the rectus femoris
  Interventions: Other: ultrasound measurement of the cross-sectional area of the rectus femoris

INTERVENTIONS:
Other: ultrasound measurement of the cross-sectional area of the rectus femoris — ultrasound measurement of the cross-sectional area of the rectus femoris at D-1 and D+3, +7 , +14

SUMMARY:
In France, the profile of patients receiving lung transplants has changed in recent years, mainly due to the advent of treatment for cystic fibrosis. This progress has led to an evolution in the patient profile, with an increase in cases of pulmonary fibrosis or COPD, and an increase in the average age of patients. In these older patients, sarcopenia, a condition characterized by loss of muscle mass, is a major concern, as it exacerbates morbidity and mortality.

After transplantation, patients are at risk of developing neuromyopathy due to their hospitalization in intensive care. There is currently no effective preventive treatment for this condition, underlining the need for early rehabilitation strategies. The combination of sarcopenia and neuromyopathy diminishes their functional capabilities on discharge from the ICU.

Muscle ultrasound, a simple, non-invasive technique, is already used to assess muscle function in intensive care patients. This study aims to evaluate the use of ultrasound to measure muscle loss in lung transplant patients, in particular by examining the rectus femoris muscle. Objectives include observing variations in the surface area of the rectus femoris muscle before and after transplantation, identifying factors influencing this variation, and exploring its relationship with post-transplant morbidity.

In summary, this study seeks to better understand muscle loss in lung transplant patients using ultrasound, in order to identify risk factors and guide the development of post-transplant rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18
* Patient registered on the lung transplant list at Hôpital Foch for a single or double-lung transplant
* Patient who did not object to inclusion in the study
* Patient affiliated to a French health insurance plan

Exclusion Criteria:

* Patient listed for a combined transplant (heart-lung, liver-lung, lung-kidney)
* Patient on national priority list (super-emergency)
* Pregnant or breast-feeding patient
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant patients at Hôpital Foch
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of the change at D7 in the cross-sectional area of the rectus femoris following lung transplantation | Baseline and Day 7

SECONDARY OUTCOMES:
Measure change in cross-sectional area of the rectus femoris at D7 according to LT pattern | Baseline and day 14
Evaluate the relationship between length of stay in intensive care unit and variation in cross-sectional area of the rectus femoris at D7 | Baseline and day 7
Determine the relationship between cross-sectional area of the rectus femoris at D-1 and Body Mass Index | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Reffienna, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, Hauts de seine, France

IPD SHARING:
Plan to Share IPD: Undecided